CLINICAL TRIAL: NCT00973648
Title: Exploring Voluntary Control of Tinnitus: A Pilot Study
Brief Title: Exploring Voluntary Control of Tinnitus
Status: Completed | Type: Observational
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Principal Investigator, Jay F. Piccirillo, MD, Professor of Otolaryngology, Director of Clinical Outcomes Research Office, Washington University School of Medicine
Other Study IDs: 09-0481
Record Dates: First submitted 2009-09-08; First posted 2009-09-09 (Estimated); Last update posted 2013-06-11 (Estimated); Status verified 2013-06

CONDITIONS: Tinnitus
Keywords: Tinnitus; Ringing in ears; Functional connectivity MRI; Voluntary control of tinnitus
MeSH Terms: conditions — Tinnitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
This pilot study aims to increase the understanding of tinnitus through the identification of potentially altered brain networks in patients who are able to voluntarily control or alter their tinnitus. Upon completion of this study, new knowledge will be gained about the changes in brain activity in people who are able to modify their tinnitus.

DETAILED DESCRIPTION:
Certain patients report that they are able to modulate the loudness or pitch of their tinnitus temporarily through various means, including attention re-direction or somatosensory mechanisms such as oral facial movements or head turn. This subset of patients may represent a unique opportunity for the researcher to gain insight into the mechanisms responsible for tinnitus.

Neural activity in the brain has been linked to increases in blood flow and blood oxygenation. These changes in the concentration of oxyhemoglobin versus deoxyhemoglobin alter the magnetic resonance signal of blood which may then be detected using an appropriate MR pulse sequence as blood-oxygen-level-dependent (BOLD) contrast. In addition to increases in blood flow due to evoked neural activity, the brain exhibits continuous low frequency spontaneous activity. These fluctuations tend to be synchronous in functionally related, but spatially distinct, regions of the brain even when not performing a prescribed task. The phrase functional connectivity has been used to implicate the neural activity that facilitates the coordinated activity of functionally related brain regions.

This study will use functional connectivity magnetic resonance imaging (fcMRI) to measure the network of synchronous brain activity in patients with tinnitus. Several targeted networks are those linked to the auditory system, attention, and control systems and the emotion systems linked to prefrontal cortex. Previously, functional MRI (fMRI) used changes in blood flow and blood oxygenation within the brain to detect which isolated regions of the brain were active during a task. The goal of functional connectivity research is to describe a pattern of interactions or a picture of the connectivity that occurs within distinct regions of the brain when the individual is not involved in a task.

ELIGIBILITY:
Inclusion Criteria:

* Adults, between the ages of 18 and 80 years.
* Idiopathic, subjective, troublesome, unilateral or bilateral, non-pulsatile tinnitus of 6 month's duration or greater.
* Patient has some voluntary control over their tinnitus, whether through attention redirection or somatosensory control, such as orofacial movements or head turn.
* Able to give informed consent.
* English-speaking.

Exclusion Criteria:

* Patients with tinnitus related to cochlear implantation, retrocochlear lesion, or other known anatomic/structural lesions of the ear and temporal bone.
* Patients with hyperacusis or misophonia (hyper-sensitivity to loud noises).
* Patients with cardiac pacemakers, intracardiac lines, implanted medication pumps, implanted electrodes in the brain, or other intracranial metal objects with the exception of dental fillings or any other contraindication for MRI scan.
* Patients with an acute or unstable medical condition including all individuals with any significant heart disease, history of seizures, pneumonia, recent hip fracture (within 3 months), acute GI bleed, uncontrolled hypertension, or other disorders which would require stabilization prior to initiation of imaging.
* Patients with a history of a brain-related injury or brain-related illness such as increased intracranial pressure, brain mass, Huntington's chorea).
* Patients currently taking psychoactive drugs that cannot be suspended for several days prior to imaging.
* Weight over 350 pounds.
* Patients with a history of claustrophobia.
* Patients who have an inability to lay flat for 1 hour.
* Patients with tinnitus related to Workman's Compensation claim or litigation-related event.
* Patients whose ability to give informed consent is in question.
* Any exclusions from radiology screening.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Speciality clinic Community health centers Solicitation of participants from American Tinnitus Association and Acoustic Neuroma Society Research database
Sampling Method: Non-Probability Sample
Enrollment: 17 (Actual)
Dates: Start 2009-08; Primary Completion 2010-08 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Changes in brain neural activity between before and after tinnitus modulation as detected on functional connectivity MRI. | After completion of functional connectivity MRI

CONTACTS AND LOCATIONS:
Overall Officials: Jay F Piccirillo, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

REFERENCES:
- [Result] Lee MH, Solowski N, Wineland A, Okuyemi O, Nicklaus J, Kallogjeri D, Piccirillo JF, Burton H. Functional connectivity during modulation of tinnitus with orofacial maneuvers. Otolaryngol Head Neck Surg. 2012 Oct;147(4):757-62. doi: 10.1177/0194599812450680. Epub 2012 Jun 6. PMID 22675003